CLINICAL TRIAL: NCT01993381
Title: Evaluation of Predictive Risk Factors of Chemotherapy-induced Nausea and Vomiting(CINV)
Brief Title: Evaluation of Predictive Risk Factors of Chemotherapy-induced Nausea and Vomiting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Byoungyong Shim, Associate professor, The Catholic University of Korea
Other Study IDs: CINV_CUKorea
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: chemotherapy-induced nausea and vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CINV of FOLFOX, FOLFIRI: moderate emetogenic chemotherapy

SUMMARY:
The most common toxicity of chemotherapy is nausea and vomiting, and appropriate management of these toxicities can help patients improve tolerance for chemotherapy. Anti-emetics including dopamine antagonist, serotonin antagonist, and substance P antagonist administered to patients according to emetogenic risk of chemotherapeutic drugs. However, patients don't always experience same nausea and vomiting for the same drugs. Therefore, it is important to determine the biomarker to predict chemotherapy-induced nausea and vomiting. Some biomarkers studies were done during the chemotherapy. However it is not definite evidence of relations between biomarkers and chemotherapy. We will hope to find any predictive biomarker of CINV.

DETAILED DESCRIPTION:
1. Primary Objective To evaluate the role of some predictive biomarkers for chemotherapy-induced nausea and vomiting
2. Secondary Objective To evaluate the clinical characteristics related to chemotherapy-induced nausea and vomiting in Korean patients
3. Study design

   Chemotherapy Day Day1 Day3 Day15

   Chemotherapy 1st cycle FOLFOX/ FOLFIRI 2nd cycle FOLFOX/ FOLFIRI Blood Sampling 1st sampling (8 a.m.) 2nd sampling (8 a.m.) 3rd sampling (8 a.m.) Evaluation of nausea and vomiting Patient's Diary (Day 1-4)
4. Evaluation of chemotherapy-induced nausea and vomiting

   * Patient's Diary consisting of the following three elements:

     1. NCI-CTCAE (National cancer institute-common toxicity criteria adverse event) version 4.0
     2. 100mm Visual Analog Scale (VAS)
     3. Functional living index- emesis
   * Patients should write 'Patient's Diary' from chemotherapy day 1 to chemotherapy day 4.
5. Evaluation of the serum levels of Biomarkers (substance P et. al.) 1) Blood sampling

   * Sample 1: 1st cycle, chemotherapy starting day 1, fasting 8 a.m.
   * Sample 2: 1st cycle, chemotherapy day 3, fasting 8 a.m.
   * Sample 3: 2nd cycle, chemotherapy starting day 1 (day 15 after 1st cycle chemotherapy), fasting 8 a.m.

     2) ELISA test for biomarkers (Sample 1,2,3)

5. Visiting Schedule

Screening Chemotherapy Time of Visit D-3 to -1 1st day of 1st cycle (Day 1) 3rd day of 1st cycle (Day 3) 4th day of 1st cycle (Day4) 1st day of 2nd cycle (Day 15) Inclusion/exclusion criteria x Informed consent x Distribution of patient's diary x Blood sampling x x x Return of patient's diary x

6. Statistical methods and data analysis Continuous variables, including serum levels of biomarkers, are expressed as median, minimum, and maximum values. Comparisons of continuous variables are made using the Mann-Whitney U test and the Kruskal-Wallis test. The chi-square test is used for comparisons of categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Histologically proven solid organ cancer
* Eastern Cooperative Oncology Group Performance status 0-2
* More than 3 months for life expectancy
* Patients scheduled to receive the first line, first cycle FOLFOX (5-FU, Oxaliplatin, Leucovorin) or FOLFIRI (5-FU, Irinotecan, Leucovorin) chemotherapy
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients who have nausea and vomiting caused by other reasons such as CNS metastases or gastrointestinal obstruction
* Patients who were exposed previously to any chemotherapy except adjuvant FL (5-FU and leucovorin)
* Patients who take anti-emetic drugs or dopamine antagonist within 72 hours prior to administration of chemotherapy
* Patients who take other drugs that may affect serum level of biomarkers (ex. steroid, megesterol, hormone replacement therapy, parenteral nutrition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to receive the first line, first cycle FOLFOX (5-FU, Oxaliplatin, Leucovorin) or FOLFIRI (5-FU, Irinotecan, Leucovorin) chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of some predictive biomarkers for chemotherapy-induced nausea and vomiting | 2 weeks after chemotherapy
  Chemotherapy Day Day1 Day3 Day15
  Chemotherapy
  1. st cycle FOLFOX/ FOLFIRI
  2. nd cycle FOLFOX/ FOLFIRI Blood Sampling 1st sampling (8 a.m.) 2nd sampling (8 a.m.) 3rd sampling (8 a.m.) Evaluation of nausea and vomiting Patient's Diary (Day 1-4)

SECONDARY OUTCOMES:
To evaluate the clinical characteristics related to chemotherapy-induced nausea and vomiting in Korean patients | 2 weeks after chemotherapy
  Patient's Diary consisting of the following three elements:
  1. NCI-CTCAE (National cancer institute-common toxicity criteria adverse event) version 4.0
  2. 100mm Visual Analog Scale (VAS)
  3. Functional living index- emesis
     * Patients should write 'Patient's Diary' from chemotherapy day 1 to chemotherapy day 4.
     * Evaluate about clinical history of patients

CONTACTS AND LOCATIONS:
Overall Officials: Byoungyong Shim, M.D., Ph.D., Principal Investigator — Department of medical oncology, The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided